CLINICAL TRIAL: NCT03778086
Title: Iridocorneal Angle and Anterior Segment Structure in Pediatric Cataract
Brief Title: Iridocorneal Angle and Anterior Segment Structure in Eyes of Children With Cataract
Acronym: ACA
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Director of Cataract Department, Wenzhou Medical University
Other Study IDs: ACA_LZL_HZ
Record Dates: First submitted 2018-12-06; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Congenital Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cataractous eyes: eyes of children with unilateral or bilateral cataract
  Interventions: Procedure: gonioscopy
- fellow eyes: fellow eyes of children with unilateral cataract
  Interventions: Procedure: gonioscopy

INTERVENTIONS:
Procedure: gonioscopy — gonioscopic observation and grading of iridocorneal angle

SUMMARY:
The aim of this study is to evaluate the morphology of iridocorneal angle and anterior segment structure in children with cataract, and to explore potential preoperative structural clues for postoperative glaucoma. The investigators included children with cataract planning to have cataract surgery in our institute. For analysis, one eye was randomly selected in a case of bilateral cataract via a random table, forming the "bilateral cataract" group; the cataractous eyes in cases of unilateral cataract composed the "unilateral cataract" group and the fellow non-cataractous eyes made up the "control" group. Exclusion criteria were: a history of ocular trauma, a history of intraocular surgery, preoperative glaucoma, steroid use before surgery, a history of maternal rubella syndrome, chronic anterior uveitis, persistent fetal vasculature, ocular anomalies associated with an increased risk of glaucoma, unable to complete examinations. The investigators recorded age at surgery, gender and relevant ocular and systemic histories. All patients underwent slit lamp biomicroscopy, dilated fundus examination and cycloplegic retinoscopy. In patients with good cooperation, The investigators obtained the axial length (AL) using IOL-Master 500 and the intraocular pressure (IOP) with a non-contact tonometer. In young patients with poor cooperation, the investigators measured the AL with a contact A-scan, the central corneal thickness (CCD) value with a handheld pachymeter and the IOP using a handheld tonometer under sedation. With a contact A-scan, the AL measurement was repeated 10 times by the same examiner and the mean value was analyzed. Corneal diameter was measured with a caliper in the operating room before cataract surgery. Under general anesthesia, a pediatric surgeon (YEZ) evaluated the iridocorneal angle with an indirect goniolens under the operating microscope. A gentle tilting of the goniolens was allowed to obtain a better view of the angle. Another experienced pediatric ophthalmologist (DDW) double checked the video recordings and graded the details of iridocorneal angle according to the Shaffer and Spaeth classification system and standard methods reported. The angle width was defined as follows: grade 0, a closed angle without visible angle structures; grade 1, a very narrow angle with Schwalbe's line visible only; grade 2, a moderately narrow angle with Schwalbe's line and trabecular meshwork visible; grade 3, an open angle with trabecular meshwork and scleral spur visible; grade 4, the widest angle with ciliary body band (CBB) visible. The iris insertion and pigmentation of the posterior trabecular meshwork were classified according to the Spaeth classification system. The iris insertion was defined as follows: A, anterior to Schwalbe's line; B, between Schwalbe's line and scleral spur; C, scleral spur visible; D, deep with ciliary body visible; E, extremely deep with > 1 mm ciliary body band. The pigmentation of trabecular meshwork was defined as follows: 0, no pigment; 1, minimal pigment; 2, mild pigment; 3, moderate pigment; 4, intense pigment. The number of iris process was defined as follows: 0, none; 1, minimal; 2, moderate; 3, marked. The width of CBB was graded according to the classification proposed by Tawara et al and defined as follows: invisible, the CBB could not be seen at all; very narrow, the CBB was narrower than the scleral spur; normal, the CBB was wider than the scleral spur. The normality of variables was tested using Kolmogorov-Smirnov test. Continuous variables are presented as mean±standard deviation or median (interquartile range) based on the normality of variables, and categorical variables are presented as frequencies and percentages. One-way ANOVA or Kruskal-Wallis test was used for overall comparison, and Dunnett test or Kruskal-Wallis One-way ANOVA was used for paired-comparison of variables between groups where appropriate. Mann-Whitney test was used for further subgroup comparison. A P value less than 0.05 was considered statistically significant. All statistical analyses were performed using SPSS version 21.0 (SPSS Inc, Chicago, Illinois, USA).

ELIGIBILITY:
Inclusion Criteria:

* children with cataract

Exclusion Criteria:

* a history of ocular trauma
* a history of intraocular surgery
* preoperative glaucoma
* steroid use before surgery
* a history of maternal rubella syndrome
* chronic anterior uveitis
* persistent fetal vasculature
* ocular anomalies associated with an increased risk of glaucoma
* unable to complete examinations.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants included eyes of children with unilateral or bilateral cataract.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Width of angle | 2016-06-01 to 2018-06-01
  The angle width was defined as follows: grade 0, a closed angle without visible angle structures; grade 1, a very narrow angle with Schwalbe's line visible only; grade 2, a moderately narrow angle with Schwalbe's line and trabecular meshwork visible; grade 3, an open angle with trabecular meshwork and scleral spur visible; grade 4, the widest angle with ciliary body band (CBB) visible

SECONDARY OUTCOMES:
Width of ciliary body band | 2016-06-01 to 2018-06-01
  The width of ciliary body band(CBB) is defined as follows: invisible, the CBB could not be seen at all; very narrow, the CBB is narrower than the scleral spur; normal, the CBB is wider than the scleral spur
The number of iris processes | 2016-06-01 to 2018-06-01
  The number of iris process is defined as follows: 0, none; 1, minimal; 2, moderate; 3, marked
Trabecular meshwork pigmentation | 2016-06-01 to 2018-06-01
  The pigmentation of trabecular meshwork is defined as follows: 0, no pigment; 1, minimal pigment; 2, mild pigment

IPD SHARING:
Plan to Share IPD: Undecided